CLINICAL TRIAL: NCT05229705
Title: The Effects of Exercise on Cognition and Brain Health in Older Adults at Risk for Type 2 Diabetes
Brief Title: Exercise in Older Adults at Risk for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Lindsay Nagamatsu, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 120336
Record Dates: First submitted 2021-12-15; First posted 2022-02-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Change
Keywords: resistance exercise; cognition; brain health; older adults; diabetes; obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Experimental group versus control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and accessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise (Experimental): Exercises will be completed in Kevin Shoemaker's (Co-I) exercise lab in the Health Sciences Building. Participants will use the programmable weight machines along with free weights to target the primary muscle groups. In addition, they will complete mini-squats, mini-lunges, and lunge walks. Participants will complete two sets of 6-8 reps. Training stimulus will be increased using the 7RM method - when 2 sets of 6-8 reps are completed with proper form and without discomfort. We will record the number of sets completed and the load lifted for each exercise for each participant at every class.
  Interventions: Behavioral: Resistance exercise
- Control (balance and tone exercise) (No Intervention): Exercises will be completed in the Health Science Exercise lab. These will include stretching exercises, range of motion exercises, basic core-strength exercises, balance exercises, and relaxation techniques. Only bodyweight will be applied (i.e., no additional loading). This group controls for confounding variables such as physical training received by traveling to the training centres, social interaction, and changes in lifestyle secondary to study participation (Liu-Ambrose et al., 2010; Liu-Ambrose et al., 2012; Nagamatsu et al., 2012; Nagamatsu et al., 2013).

INTERVENTIONS:
Behavioral: Resistance exercise — Participants in this exercise group will receive progressive resistance training.
  Arms: Resistance exercise

SUMMARY:
Older adults with type 2 diabetes experience neurocognitive decline and are at higher risk for developing dementia. Consequently, older adults at-risk for developing type 2 diabetes (i.e., those who are overweight and/or prediabetic) are at higher risk for neurocognitive decline, and intervening at this point may prevent or delay the onset of such decline. One promising lifestyle intervention that has been shown to improve cognitive function and brain health in other populations is resistance exercise. We previously conducted a 6-month resistance training randomized controlled trial (RCT) pilot study that showed a large scale trial would be viable and feasible. Consequently, we would like to explore resistance exercise as a lifestyle intervention to improve cognition and brain structure in older adults at risk for diabetes.

DETAILED DESCRIPTION:
The effects of exercise on cognition and brain structure in older adults at risk for type 2 diabetes: A 3T MRI study

Objectives/research questions:

In this study the research questions included:

1. Does twice-weekly resistance training impact cognitive function compared to balance-and-tone exercises in older adults at risk for diabetes?
2. Can resistance training modify brain structure and volume in various brain structures, particularly the hippocampus, compared with balance-and-tone training (control) in older adults at risk for diabetes?

Hypotheses:

1. 6-months of resistance training will improve cognitive function in older adults at risk for diabetes compared to balance and tone training. We predict to see significant improvements in executive function in the resistance-trained group compared with the balance-and-tone group.
2. 6-months of resistance training will preserve hippocampal structure and volume in older adults at risk for diabetes compared to balance-and-tone exercises.

Design:

6-month Randomized Controlled Trial, Single Blinded Study Arms: 1) Experimental: Resistance Training (RT) 2) Control: Balance-and-Tone (BAT) Training

Methodology:

Screening: Participants will complete the initial screening over the phone. Interested participants will be sent the Letter of Information (via e-mail, or preferred method) to get more detailed information about the study. Those who are eligible will be scheduled to come into the lab for baseline assessments.

Baseline assessments: The following questionnaires/tests/assessments will be completed. Participants can decline any or all the tests or can choose to not answer any of the questions. If they choose to not answer a question or complete a test that is necessary for confirming eligibility, they will be excluded from the rest of the study.

Randomization: Once participants complete all baseline assessments, they will be randomly assigned to one of two groups using a random number generator. All participants have equal chances of getting into the 2 groups.

Total time to complete baseline assessments in the lab (excluding magnetic resonance imaging; MRI) will be 2 to 2.5 hours.

1. Basic demographic questionnaire: Will be used to characterize our sample.
2. Functional Comorbidity Index (FCI): An 18-item list of diagnoses used to determine comorbidities.
3. Sleep questionnaire: Determines quality and quantity of sleep over a one-month time span and the previous night specifically.
4. Activities-Specific Balance Scale (ABC): A 16-item self-report questionnaire used to assess balance and functional mobility. Participants rate their balance confidence in their ability to perform daily activities.
5. The Lawton Instrumental Activities of Daily Living (IADL): A self-report questionnaire used to assess independent living skills.
6. Physical Activity Scale for the Elderly (PASE): Used to measure the level of self-reported physical activity, and consists of 12 questions about leisure, household, and work-related daily activity.
7. The Canadian Diabetes Risk Questionnaire (CANRISK): A 12-item self-report questionnaire used to determine if participants are at high-risk of having pre-diabetes or type II diabetes.
8. Diabetes questionnaire: A questionnaire to determine risk of diabetes.
9. Geriatric Depression scale: A 15-item questionnaire used to test for the presence of depression. If depression is suspected, the Primary Investigator (PI) will ensure that the participant is provided with a copy of the questionnaire and will advise the participant to make an appointment with their family physician to discuss the results.
10. 12-Item Short Form Survey (SF-12): Self-reported survey of health.
11. Six-minute walk test: Used to assess aerobic fitness. Participants walk at their usual speed for a total of 6 minutes in the hallway outside of our lab. The total distance walked in meters is recorded.
12. Timed Up and Go test (TUG): Used to assess mobility. Participants are seated in a chair and must stand up, walk a distance of 3 meters at their usual pace, turn around, return to their chair, and sit back down. The time to complete each of two separate trials is recorded in seconds.
13. Short Physical Performance Battery (SPPB): Used to assess gait speed, balance, and lower extremity physical function using tasks that mimic daily activities; includes three tasks: Standing Balance Task, Walking Speed Task, and Chair Stand Test.
14. Falls history: Used to assess mobility and falls-risk.
15. One-repetition maximum (1RM): A physical measure of an individual's maximum muscle strength during a single repetition and is used to determine the desired load for resistance training. Exercise includes leg press, latissimus pulldown, leg curl, chest press, bicep curls, tricep extensions, and pulley rows.
16. Paired Associative Learning (PAL) Touchscreen Task: Used to test learning and remembering of three objects that are associated with a correct spatial location on the screen.
17. Trail Unique-Non-Matching-Location (TUNL) Task: This is a working spatial memory task that involves selecting a different stimulus (non-matching) to the stimulus presented on the screen after a delay period. The stimuli are presented in locations far apart or close together to challenge spatial memory.
18. Progressive Ratio (PR) Touchscreen Task: This task tests motivation and attention and involves repeatedly touching a square stimulus at the center of the screen for points in a single trial. The number of touches required for points increases on a ramp scale, which begins at one touch and then is increased by four on each subsequent trial. If the participant stops responding for 5 minutes, the task stops, and the point of break (stopping) is recorded.
19. Mini-Mental Status Examination (MMSE): Used as a screening tool for cognitive impairment. This 11-item test assesses global cognitive function in the domains of orientation, registration, attention and calculation, recall, and language. Maximum score is 30.
20. Montreal Cognitive Assessment (MoCA): Used as a screening tool for mild cognitive impairment. This test assesses cognitive ability in the domains of attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Maximum score is 30.
21. Alzheimer's Disease Assessment Scale Cognitive Subscale 11 (ADAS-Cog-11): Test with 11 tasks measuring various cognitive functions (memory, language, praxis, attention). Used widely in clinical trials to assess cognitive dysfunction and Alzheimer's Disease.
22. Trail Making Test (TMT): Used to assess executive function in the areas of visual attention (Part A) and set-shifting (the ability to shift attention between one task and another; Part B). The time to complete this test is recorded in seconds.
23. Stroop: Used to assess executive function in the areas of selective attention, processing speed, and cognitive flexibility. The time to complete this test is recorded in seconds.
24. Digit Span: Used to assess working memory. Participants are required to memorize and recall a series of number lists both forward and backward.
25. Blood Tests: We will collect blood samples to test glycated hemoglobin and fasting glucose levels to determine diabetes status (pre-diabetes, diabetes) and biomarkers of brain health (brain-derived neurotrophic factor, insulin-like growth factor 1). Blood will be drawn in the exercise health lab. Blood draws will be done by registered nurse (RN) Arlene Fleischhauer in Co-investigator (Co-I) Kevin Shoemaker's lab or by our trained research student, Olivia Ghosh-Swaby.
26. Physical Activity Readiness Questionnaire (PAR-Q): The researchers will provide this form to be filled out by their family physician and returned. The form outlines the exercise program in the study to the family physician so they can advise appropriately.

MRI Screening form: Used to screen for eligibility for MRI scanning. MRI scanning will be done at the Centre for Functional and Metabolic Mapping at the Robarts Research Institute.

The one-hour scan will consist of the following:

1. Structural MRI 3Tesla (3T) scan (T1) to examine brain structure images to subject-specific structural images.
2. Resting-state functional connectivity to examine activation in the resting state network.

Exercise intervention: Exercise classes will run two times per week for 26 weeks (6 months). Classes will be group classes, with up to 5 participants in each class. All classes will be 1 hour total - 10 minutes warm up, 40 minutes main exercises, 10 minutes cool-down. Class leaders will be present during all classes to monitor participants for shortness of breath, proper technique, and to reduce any risks/hazards during the exercise classes. This protocol has been used extensively by the PI (Liu-Ambrose et al., 2010; Liu-Ambrose et al., 2012; Nagamatsu et al., 2012; Nagamatsu et al., 2013).

RESISTANCE TRAINING: Exercises will be completed in Kevin Shoemaker's exercise lab in the Health Sciences Building. Participants will use the programmable weight machines along with free weights to target primary muscle groups. In addition, they will complete mini-squats, mini-lunges, and lunge walks. Participants will complete two sets of 6-8 reps. Training stimulus will be increased using the "7-RM" method - when 2 sets of 6-8 reps are completed with proper form and without discomfort. We will record the number of sets completed and the load lifted for each exercise for each participant at every class.

BALANCE AND TONE (Control): Exercises will be completed in the Health Science Exercise lab (same as above). These will include stretching exercises, range of motion exercises, basic core-strength exercises, balance exercises, and relaxation techniques. Only bodyweight will be applied (i.e., no additional loading). This group controls for confounding variables such as physical training received by traveling to the training centres, social interaction, and changes in lifestyle secondary to study participation

Compliance: Class attendance will be recorded by class instructors.

Adverse events: All adverse events that occur during exercise classes will be recorded and reported immediately.

Fidelity Questionnaire: To ensure consistency across exercise classes and help identify any potential program issues, a questionnaire was completed by a nonstudy affiliate once per month, where he/she attended and evaluated a randomly selected RT and BAT session.

Monthly assessments: During the 6-month exercise intervention, participants will complete the following assessments monthly.

1. PASE
2. Falls calendar

Final assessments: All baseline assessments will be completed at trial completion (26 weeks) INCLUDING MRI scanning and blood draw with consent.

Significance:

This study will elucidate whether resistance exercise is a plausible intervention for cognitive decline in those at risk for diabetes. The findings of this study will also determine a viable time point to intervene before the onset of a significant decline in older adults with disrupted metabolic homeostasis. Additionally, this study has the potential to identify cost-effective and accessible strategies to improve cognitive function in those at-risk for decline. Given the enormous burden (financial, quality of life, independence) of cognitive decline in our aging society, the potential positive implications of our study cannot be overstated.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling
2. Aged 60-80 years
3. "At-risk" for diabetes, where they have one of the following: i) blood glucose level of 6.1-7 mmol/L, ii) body mass index > 25, or iii) score > 21 on the CANRISK diabetes questionnaire
4. Score > 24/30 on MMSE
5. Score > 6/8 on the IADL scale
6. Visual acuity of at least 20/40, with or without corrective lenses
7. Speak and understand English fluently
8. Complete the PAR-Q
9. Obtain physician's clearance to start a supervised exercise program

Exclusion Criteria:

1. Current medical condition for which exercise is contraindicated
2. Participated regularly in resistance or aerobic training in the last 6 months
3. Diagnosed with neurodegenerative disease (including dementia, Alzheimer's disease, or Parkinson's disease)
4. Experienced a vascular incident (e.g., stroke, myocardial infarction)
5. Diagnosed with a psychiatric condition
6. Untreated depression and scored 5 or less on the Geriatric Depression Scale
7. Currently on hormone replacement therapy
8. Clinically significant peripheral neuropathy or severe musculoskeletal or joint disease
9. Currently taking psychotropic medications
10. Cannot blood draw

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Trail Making Test | 5 minutes
  Used to assess executive function in the areas of visual attention (Part A) and set-shifting (the ability to shift attention between one task and another; Part B). The time to complete this test is recorded in seconds.

SECONDARY OUTCOMES:
Paired Associative Learning (PAL) Touchscreen Task | 20 minutes
  Used to test learning and remembering of three objects that are associated with a correct spatial location on the screen.
Trail Unique-Non-Matching-Location (TUNL) Task | 20 minutes
  This is a working spatial memory task that involves selecting a different stimulus (non-matching) to the stimulus presented on the screen after a delay period. The stimuli are presented in locations far apart or close together to challenge spatial memory.
Progressive Ratio (PR) Touchscreen Task | 20 minutes
  This task tests motivation and attention. The task involves touching a square stimulus at the center of the screen repeatedly for points in a single trial. The number of touches required for points increases on a ramp scale, which begins at one touch for points and then is increased by four on each subsequent trial for points. If the participant stops responding for 5 minutes, the task stops, and the point of break (stopping) is recorded.
Stroop Test | 5-10 minutes
  Used to assess executive function in the areas of selective attention, processing speed, and cognitive flexibility. The time to complete this test is recorded in seconds.
Digit Span Test | 5-10 minutes
  Used to assess working memory. Participants are required to memorize and recall a series of number lists both forward and backward.
Alzheimer's Disease Assessment Scale Cognitive Subscale 11 | 15 minutes
  Test with 11 tasks measuring various cognitive functions (memory, language, praxis, attention). Used widely in clinical trials to assess cognitive dysfunction and Alzheimer's Disease.
Glycated hemoglobin A1c (HbA1C) | 5-10 minutes
  We will collect blood samples to test glycated hemoglobin levels to determine diabetes status (pre-diabetes, diabetes). Blood will be drawn from a cubital vein into a 7.5 ml tube. Blood draws will be done by RN Arlene Fleischhauer in Co-I Kevin Shoemaker's lab or by trained support staff, Olivia Ghosh-Swaby.
Fasting plasma glucose | 5-10 minutes
  We will collected via a glucometer finger prick
Height | 5 minutes
  Measured in m; used to calculate body mass index (kg/m^2)
Weight | 5 minutes
  Measured in kg; used to calculate body mass index (kg/m^2)
Triglyceride levels | 30 minutes
  Will be assessed via serum samples measured by ELISA.
Inflammatory markers | 30 minutes
  Will be assessed via serum samples measured by ELISA.
Brain-derived neurotrophic factor levels | 1 hour
  Will be assessed via serum samples measured by ELISA.
Insulin-like growth factor levels | 1 hour
  Will be assessed via serum samples measured by ELISA.
One repetition maximum | 10-15 minutes
  One-repetition maximum is a physical measure of an individual's maximum muscle strength during a single repetition and is used to determine the desired load for resistance training.
Six-minute walk test | 6 minutes
  Used to assess aerobic fitness. Participants walk at their usual speed for a total of 6 minutes in the hallway outside of our lab. The total distance walked in meters is recorded.
Short Physical Performance Battery (SPPB) - Task 1 | 5 minutes
  Used to assess gait speed, balance, and lower extremity physical function using tasks that mimic daily activities; the Standing Balance Task requires participants to stand unassisted (side-by-side standing, semi-tandem standing, and tandem standing) for a period of 10 seconds each; scored in conjunction with SPPB Tasks 2 & 3 to produce one final SPPB score
Short Physical Performance Battery (SPPB) - Task 2 | 5 minutes
  Used to assess gait speed, balance, and lower extremity physical function using tasks that mimic daily activities; the Walking Speed Task requires participants to walk 4 metres at their usual pace; measured in seconds; scored in conjunction with SPPB Tasks 1 & 3 to produce one final SPPB score
Short Physical Performance Battery (SPPB) - Task 3 | 5 minutes
  Used to assess gait speed, balance, and lower extremity physical function using tasks that mimic daily activities; the Chair Stand Test requires participants to stand up from a chair 5 times consecutively (without the use of their arms if possible); measured in seconds; scored in conjunction with SPPB Tasks 1 & 2 to produce one final SPPB score
Timed Up and Go Test | 5-10 minutes
  Used to assess mobility. Participants are seated in a chair and must stand up, walk a distance of 3 meters at their usual pace, turn around, return to their chair, and sit back down. The time to complete each of two separate trials is recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Nagamatsu, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furlano JA, Nagamatsu LS. Feasibility of a 26-Week Exercise Program to Improve Brain Health in Older Adults at Risk for Type 2 Diabetes: A Pilot Study. Can J Diabetes. 2021 Aug;45(6):546-552. doi: 10.1016/j.jcjd.2020.11.001. Epub 2020 Nov 13. PMID 33358932
- [Background] Liu-Ambrose T, Nagamatsu LS, Graf P, Beattie BL, Ashe MC, Handy TC. Resistance training and executive functions: a 12-month randomized controlled trial. Arch Intern Med. 2010 Jan 25;170(2):170-8. doi: 10.1001/archinternmed.2009.494. PMID 20101012
- [Background] Nagamatsu LS, Handy TC, Hsu CL, Voss M, Liu-Ambrose T. Resistance training promotes cognitive and functional brain plasticity in seniors with probable mild cognitive impairment. Arch Intern Med. 2012 Apr 23;172(8):666-8. doi: 10.1001/archinternmed.2012.379. No abstract available. PMID 22529236
- [Background] Awad N, Gagnon M, Messier C. The relationship between impaired glucose tolerance, type 2 diabetes, and cognitive function. J Clin Exp Neuropsychol. 2004 Nov;26(8):1044-80. doi: 10.1080/13803390490514875. PMID 15590460